CLINICAL TRIAL: NCT02536508
Title: A Randomized, Double-Blind, Parallel-Group, 52-Week, Chronic-Dosing, Multi-Center Study to Assess the Safety and Tolerability of PT010, PT009 and PT003 in Subjects With Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Brief Title: Study to Assess the Safety and Tolerability of PT010, PT009 and PT003 in Subjects With Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT010008; NCT03313570 (obsolete NCT alias)
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- BGF MDI (PT010) 320/14.4/9.6 μg (Experimental): Budesonide, Glycopyrronium, and Formoterol Fumarate (BGF) metered dose inhaler (MDI) (PT010, BGF MDI)
  Interventions: Drug: BGF MDI 320/14.4/9.6 μg
- GFF MDI (PT003) 14.4/9.6 μg (Experimental): Glycopyrronium and Formoterol Fumarate (GFF) metered dose inhaler (MDI) (PT003, GFF MDI)
  Interventions: Drug: GFF MDI 14.4/9.6 μg
- BFF MDI (PT009) 320/9.6 μg (Experimental): Budesonide and Formoterol Fumarate (BFF) metered dose inhaler (MDI) (PT009, BFF MDI)
  Interventions: Drug: BFF MDI 320/9.6 μg

INTERVENTIONS:
Drug: BGF MDI 320/14.4/9.6 μg — Budesonide, Glycopyrronium, and Formoterol Fumarate
  Other Names: BGF MDI
  Arms: BGF MDI (PT010) 320/14.4/9.6 μg
Drug: GFF MDI 14.4/9.6 μg — Glycopyrronium and Formoterol Fumarate
  Other Names: GFF MDI
  Arms: GFF MDI (PT003) 14.4/9.6 μg
Drug: BFF MDI 320/9.6 μg — Budesonide and Formoterol Fumarate
  Other Names: BFF MDI
  Arms: BFF MDI (PT009) 320/9.6 μg

SUMMARY:
Study to Assess the Safety and Tolerability of PT010, PT009 and PT003 in Subjects with Moderate to Very Severe Chronic Obstructive Pulmonary Disease

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Parallel-Group, 52-Week, Chronic-Dosing, Multi-Center Study to Assess the Safety and Tolerability of PT010, PT009 and PT003 in Subjects with Moderate to Very Severe Chronic Obstructive Pulmonary Disease

ELIGIBILITY:
Inclusion Criteria:

Given their signed written informed consent to participate. Must have agreed to participate in and complete the lead-in Study PT010006.(NCT02497001)

Exclusion Criteria:

Severe osteoporosis Unable to achieve an acceptable DEXA scan Inability to achieve pupil dilation to at least 6 mm Subjects with an implanted artificial intraocular lens or are scheduled to undergo cataract surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, Study Director — Pearl Therapeutics; Paul Dorinsky, MD, Study Director — Pearl Therapeutics
Locations (59):
- United States (59):
  - Research Site, Dothan, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Fullerton, California
  - Research Site, Gold River, California
  - Research Site, Poway, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Sacramento, California
  - Research Site, Clearwater, Florida
  - Research Site, Miami, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Dacula, Georgia
  - Research Site, Norcross, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Edina, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Woodbury, Minnesota
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Easley, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Old Point Station, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Seneca, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Johnson City, Tennessee
  - Research Site, Kingwood, Texas
  - Research Site, Longview, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Abingdon, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Singh D, Hurst JR, Martinez FJ, Rabe KF, Bafadhel M, Jenkins M, Salazar D, Dorinsky P, Darken P. Predictive modeling of COPD exacerbation rates using baseline risk factors. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107314. doi: 10.1177/17534666221107314. PMID 35815359
- See also: PT010008-01_Protocol_Version_2.0_REDACTED.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=PT010008&attachmentIdentifier=d9239f6b-90fa-4a08-94a5-e39e103a3405&fileName=PT010008-01_Protocol_Version_2.0_REDACTED.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study randomized subjects at 69 sites in the United States from September 2015 to September 2017. The entire study period was scheduled to take up to approximately 58 weeks for each individual subject from the time of screening through the follow-up period.
Pre-assignment Details: Subjects were randomized in a 2:2:1 scheme (BGF MDI:GFF MDI:BFF MDI).
Groups:
- BGF MDI 320/14.4/9.6 ug: Budesonide Gylcopyrronium and Formoterol Fumarate Inhalation Aerosol 320/14.4/9.6 ug
- GFF MDI 14.4/9.6 ug: Glycopyrronium and Formoterol Fumarate Inhalation Aerosol 14.4/9.6 ug
- BFF MDI 320/9.6 ug: Budesonide and Formoterol Fumarate Inhalation Aerosol 320/9.6 ug
Period: Overall Study
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug
Started (Safety population) | 194 | 174 | 88
Completed | 142 | 130 | 65
Not Completed | 52 | 44 | 23
Not completed — Withdrawal by Subject | 18 | 13 | 7
Not completed — Adverse Event | 14 | 13 | 6
Not completed — Lost to Follow-up | 12 | 4 | 0
Not completed — Lack of Efficacy | 3 | 5 | 4
Not completed — Protocol Discontinuation Criteria | 3 | 2 | 2
Not completed — Physician Decision | 0 | 4 | 2
Not completed — Major Protocol Deviation | 2 | 2 | 2
Not completed — Administrative Reasons | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included only subjects who signed ICF for Study PT010008 and received any amount of study drug (other than Symbicort).
Groups:
- Total: Total of all reporting groups
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug | Total
Number analyzed (Participants) | 194 | 174 | 88 | 456
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Safety Population
  Years | 62.6 (7.9) | 62.4 (7.8) | 64.0 (7.2) | 62.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Female | 92 | 87 | 35 | 214
    Male | 102 | 87 | 53 | 242
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Hispanic or Latino | 9 | 5 | 6 | 20
    Not Hispanic or Latino | 185 | 169 | 82 | 436
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Safety Population
  Participants
    Black | 13 | 17 | 9 | 39
    White | 179 | 156 | 79 | 414
    Asian | 0 | 1 | 0 | 1
    Other | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in BMD of the Lumbar Spine
Description: Percent change from baseline in BMD of the lumbar spine T-Score at Week 52.
Time Frame: at week 52
Population: BMD Population was defined as all evaluable subjects in the Safety Population who had a baseline BMD assessment and at least 1 on-treatment BMD assessment. Subjects were analyzed according to actual study drug received.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug
Number analyzed (Participants) | 128 | 123 | 57
Percentage | -0.093 [-0.739 to 0.557] | 0.379 [-0.28 to 1.042] | -0.120 [-1.087 to 0.857]

2. Primary Outcome: Change From Baseline in the LOCS III (P) Score at Week 52
Description: Change from baseline in the LOCS III (P) score (Severity of Posterior Subcapsular Cataract) at Week 52. P score is reported as a decimalized scale ranging from 0.1 (indicating a completely clear or colorless lens) to 5.9 (indicating complete opacification on the posterior capsule). A negative change in P score indicates an improvement and a positive change indicates a deterioration of LOCS III. A change in P score within 0.5 is an acceptable variation margin.
Time Frame: at week 52
Population: Ophthalmologic Population was defined as all evaluable subjects in the Safety Population who had a baseline ophthalmologic assessment and at least 1 on-treatment ophthalmologic assessment. Subjects were analyzed according to actual study drug received.
Measure: Least Squares Mean (95% Confidence Interval); unit: P-Score
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug
Number analyzed (Participants) | 132 | 125 | 54
P-Score | 0.153 [0.079 to 0.227] | .026 [-0.055 to 0.106] | 0.022 [-0.090 to 0.135]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of administration of the first dose of study drug to the time of the final follow-up telephone call. Serious Adverse events were collected from the time subject signed Informed Consent to the time of the final follow-up telephone call up to approximately 54 weeks.
Description: The Safety Population was defined as all subjects who were randomized to treatment and received at least 1 dose of the study drug.
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug
All-Cause Mortality (participants affected / at risk) | 3/194 | 1/174 | 0/88
Serious Adverse Events (participants affected / at risk) | 33/194 | 22/174 | 7/88
Other Adverse Events (participants affected / at risk) | 62/194 | 51/174 | 30/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI 320/14.4/9.6 ug (N=194) | GFF MDI 14.4/9.6 ug (N=174) | BFF MDI 320/9.6 ug (N=88)
Chronic Pulmonary Obstructive Disease (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 9 (11) | 2 (3)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave invesion (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI 320/14.4/9.6 ug (N=194) | GFF MDI 14.4/9.6 ug (N=174) | BFF MDI 320/9.6 ug (N=88)
Upper Respiratory Tract Infection (Infections and infestations) | 18 (24) | 17 (20) | 6 (6)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 9 (11) | 5 (6) | 6 (6)
Sinusitis (Infections and infestations) | 11 (14) | 6 (7) | 2 (3)
Urinary Tract Infection (Infections and infestations) | 10 (10) | 6 (9) | 4 (4)
Bronchitis (Infections and infestations) | 12 (13) | 8 (10) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 5 (5)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 9 (9) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2016-03-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT02536508/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT02536508/SAP_001.pdf